CLINICAL TRIAL: NCT03601663
Title: Exploring the Effect of an eHealth Intervention on Women's Physical Activity Behaviour
Brief Title: Exploring the Effect of an Intervention on Women's Physical Activity Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Jennifer Brunet, Associate Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: eHealth_Women_PA
Record Dates: First submitted 2018-07-04; First posted 2018-07-26 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Physical Activity
Keywords: physical activity; obesity; pilot study; randomized controlled trial; women; eHealth
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants in the main experimental group will receive a copy of the Canadian Physical Activity Guidelines that provide basic information about and recommendations for physical activity, a wearable activity tracker to support self-monitoring, and autonomy-support delivered through weekly emails to help enhance motivation for physical activity.
  Interventions: Behavioral: Physical Activity Information; Behavioral: Physical Activity Monitoring; Behavioral: Autonomy-support
- Group 2 (Active Comparator): Participants in this comparison group will receive a copy of the Canadian Physical Activity Guidelines that provide basic information about and recommendations for physical activity, and a wearable activity tracker to support self-monitoring. They will not receive any specific support to enhance motivation for physical activity.
  Interventions: Behavioral: Physical Activity Information; Behavioral: Physical Activity Monitoring
- Group 3 (Active Comparator): Participants in this information-only comparison group will receive a copy of the Canadian Physical Activity Guidelines that provide basic information about and recommendations for physical activity.
  Interventions: Behavioral: Physical Activity Information

INTERVENTIONS:
Behavioral: Physical Activity Information — Participants will receive a copy of the Canadian Physical Activity Guidelines.
Behavioral: Physical Activity Monitoring — Participants will receive a wearable activity tracker (Polar A300).
  Arms: Group 1; Group 2
Behavioral: Autonomy-support — Participants will receive eight autonomy-supportive weekly emails containing information and activities to help them set goals and make changes to become physically active.
  Arms: Group 1

SUMMARY:
Physical activity has been shown to reduce the risk of chronic diseases and promote physical and mental health and wellbeing, yet few women are active enough to see these benefits. Wearable activity trackers show promise for helping people increase their physical activity levels by supporting self-monitoring. However, few researchers have examined how providing people with these devices impacts physical activity levels, or motivation for physical activity which is a significant and robust predictor of physical activity. Based on previous research, it is possible that women's physical activity levels would be more likely to increase if they received an autonomy-supportive intervention to enhance motivation in addition to a wearable activity tracker. A pilot, three-armed randomized controlled trial was developed to test this hypothesis and to assess if changes in perceived autonomy-support, basic psychological need satisfaction/thwarting, motivational regulations, wellbeing indicators are associated with changes in physical activity over time.

ELIGIBILITY:
All participants will need to meet the following inclusion criteria to participate in the intervention:

1. Are a woman between the ages of 18 and 65 years
2. Can understand, read, and speak in English
3. Are able to safely engage in physical activity
4. Are not currently pregnant or lactating
5. Currently participating in less than 150 minutes of moderate or vigorous intensity physical activity and less than two strength training sessions per week
6. Are overweight or obese (i.e., have a body mass index greater than 25kg/m2)
7. Have access to the Internet and an email account
8. Have not used a wearable activity tracker within the past year (e.g., Fitbit, Apple Watch, Garmin, Polar)
9. Live within 50km of the University of Ottawa

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Physical activity behaviour: International Physical Activity Questionnaire Short Form (IPAQ-S) | Baseline (week 0), post-intervention (week 9), and follow-up (week 21).
  Change in self-reported physical activity (over the past 7 days) from baseline to post-intervention, and from post-intervention to follow-up.
Physical activity behaviour: Custom strength and resistance training questionnaire | Baseline (week 0), post-intervention (week 9), and follow-up (week 21).
  Change in strength and resistance training habits from baseline to post-intervention, and from post-intervention to follow-up.

SECONDARY OUTCOMES:
Physical activity behaviour: Direct measure | Duration of intervention phase (8 weeks).
  Change in weekly directly measured levels of physical activity as measured by accelerometers (Polar A300), which will be worn by participants assigned to Group 1 and Group 2 during waking hours for the duration of the intervention.
Perceived autonomy support: Perceived Autonomy Support Scale for Exercise Settings (PASSES; Hagger et al., 2007) | Baseline (week 0), post-intervention (week 9), and follow-up (week 21).
  Change in perceived autonomy support for physical activity from baseline to post-intervention, and from post-intervention to follow-up.
Basic psychological need satisfaction: Psychological Need Satisfaction in Exercise Scale (PNSE; Wilson, Rogers, Rodgers, & Wild, 2006) | Baseline (week 0), post-intervention (week 9), and follow-up (week 21).
  Change in basic psychological need satisfaction for physical activity from baseline to post-intervention, and from post-intervention to follow-up.
Motivational regulations: Behavioral Regulation in Exercise Questionnaire (BREQ-2R; Markland & Tobin, 2004; Wilson, Rodgers, Loitz, & Scime, 2006) | Baseline (week 0), post-intervention (week 9), and follow-up (week 21).
  Change in motivational regulations for physical activity from baseline to post-intervention, and from post-intervention to follow-up.
Basic psychological need thwarting: Psychological Need Thwarting Scale (PNTS; Bartholomew, Ntoumanis, Ryan, & Thøgersen-Ntoumani, 2011) | Baseline (week 0), post-intervention (week 9), and follow-up (week 21).
  Change in basic psychological need thwarting activity from baseline to post-intervention, and from post-intervention to follow-up.
Positive and Negative Affect Schedule (I-PANAS-SF; Thompson, 2016; Watson, Clark, & Tellegen, 1988). | : Baseline (week 0), post-intervention (week 9), and follow-up (week 21).
  Change in affect from baseline to post-intervention, and from post-intervention to follow-up.
Vitality: Subjective Vitality Scale (Ryan & Frederick, 1997). | Baseline (week 0), post-intervention (week 9), and follow-up (week 21).
  Change in vitality affect from baseline to post-intervention, and from post-intervention to follow-up.
Depression: Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001). | Baseline (week 0), post-intervention (week 9), and follow-up (week 21).
  Change in depressive symptoms from baseline to post-intervention, and from post-intervention to follow-up.
Wearable activity tracker usage: Multiple choice questions | Post-intervention (week 9).
  Frequency of wearable activity tracker usage in general during the intervention phase for participants randomized to Group 1 or Group 2.
Recruitment rates | Duration of recruitment and intervention phases (9 weeks).
  The number of eligible participants who enrol in the study out of the number assessed for eligibility.
Retention rates | Duration of recruitment and intervention phases (9 weeks).
  The number of participants completing all scheduled assessments.
Acceptability: Open ended questions | Duration of recruitment and intervention phases (9 weeks).
  For participants randomized to Group 1, what participants liked, disliked, and would change about the intervention.
Body mass | Baseline (week 0) and post-intervention (week 9).
  Change in body mass measured from baseline to post-intervention as determined using a scale (Tanita BWB 800S).
Body composition | Baseline (week 0) and post-intervention (week 9).
  Change in body composition from baseline to post-intervention as determined by a scale (Tanita BWB 800S) that uses bioelectrical impedance to assess body composition.
Waist circumference | Baseline (week 0) and post-intervention (week 9).
  Change in waist circumference from baseline to post-intervention as measured using a measuring tape.

OTHER OUTCOMES:
Sociodemographic questionnaire | Baseline (week 0).
  Sociodemographic and health information will be collected at baseline to describe the sample. Measures include age, marital status, race, level of education, employment status, household income, number and age of children, self-rated health, medical conditions, menstrual status, smoking history, and weight-related goals.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartholomew KJ, Ntoumanis N, Ryan RM, Thogersen-Ntoumani C. Psychological need thwarting in the sport context: assessing the darker side of athletic experience. J Sport Exerc Psychol. 2011 Feb;33(1):75-102. doi: 10.1123/jsep.33.1.75. PMID 21451172
- [Background] Hagger, M. S., Chatzisarantis, N. L., Hein, V., Pihu, M., Soós, I., & Karsai, I. (2007). The perceived autonomy support scale for exercise settings (PASSES): Development, validity, and cross-cultural invariance in young people. Psychology of Sport and Exercise, 8(5), 632-653. doi:10.1016/j.psychsport.2006.09.001
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Markland, D., & Tobin, V. (2004). A modification to the behavioural regulation in exercise questionnaire to include an assessment of amotivation. Journal of Sport & Exercise Psychology, 26, 191-196.
- [Background] Ryan RM, Frederick C. On energy, personality, and health: subjective vitality as a dynamic reflection of well-being. J Pers. 1997 Sep;65(3):529-65. doi: 10.1111/j.1467-6494.1997.tb00326.x. PMID 9327588
- [Background] Thompson, E. R. (2016). Development and validation of an internationally reliable short-form of the Positive and Negative Affect Schedule (PANAS). Journal of Cross-Cultural Psychology, 38(2), 227-242. doi:10.1177/0022022106297301
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Wilson, P. M., Rodgers, W. M., Loitz, C., & Scime, G. (2006). "It's who I am… really!" The importance of integrated regulation in exercise contexts. Journal of Applied Biobehavioural Research, 11(2), 79-104.
- [Background] Wilson, P. M., Rogers, T., Rodgers, W. M., & Wild, C. (2006). The psychological need satisfaction in exercise scale. Journal of Sport & Exercise Psychology, 28, 231-251.
- [Derived] Brunet J, Sharma S, Price J, Black M. Acceptability and Usability of a Theory-Driven Intervention via Email to Promote Physical Activity in Women Who Are Overweight or Obese: Substudy Within a Randomized Controlled Trial. JMIR Form Res. 2023 Oct 3;7:e48301. doi: 10.2196/48301. PMID 37788048
- [Derived] Black M, Brunet J. A Wearable Activity Tracker Intervention With and Without Weekly Behavioral Support Emails to Promote Physical Activity Among Women Who Are Overweight or Obese: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Dec 16;9(12):e28128. doi: 10.2196/28128. PMID 34927590